CLINICAL TRIAL: NCT05129865
Title: A Phase 1, Double Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of LYT-300 in Healthy Volunteers, and a Phase 1b/2a Study Part to Assess Effects of a Single Dose of LYT-300 vs. Placebo on the Response to a Standardized Behavioural Challenge in Healthy Volunteers
Brief Title: LYT-300 in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PureTech (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYT-300-2021-101
Record Dates: First submitted 2021-10-31; First posted 2021-11-22 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Part 1 consists of 1 Arm with crossover of active treatment and placebo; Part 2 consists of 1 Arm with active treatment; Part 3 consists of 4 Arms with active treatment or placebo; Part 4 consists of 2 arms with active or placebo.
Who Masked: Participant, Investigator
Masking Description: Parts 1, 2 and 3 are double blind during the data collection. Determination for dose escalation may be made under unblinded conditions by assessors.
  Part 4 consists of 2 groups. Group 1 (the validation group) will be single-arm placebo. Group 2 (the test group) will be double blind during data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- LYT-300 in healthy volunteers LYT-300, Doses TBD (Experimental): Subjects will crossover across 3 dosing periods in which they will receive placebo and two experimental dose levels
  Interventions: Drug: LYT-300; Other: Placebo
- LYT-300 in healthy volunteers LYT-300 (Experimental): LYT-300, Dose TBD with and without food, separated by 7-day washout
  Interventions: Drug: LYT-300
- LYT-300, Dose TBD QAM every 24 h for 7 days (Experimental)
  Interventions: Drug: LYT-300
- Placebo QAM every 24 h for 7 days (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo QHS every 24 h for 7 days (Placebo Comparator)
  Interventions: Drug: LYT-300; Other: Placebo
- LYT-300 in healthy volunteers LYT-300, Dose TBD QHS every 24 h for 7 days (Experimental)
  Interventions: Drug: LYT-300; Other: Placebo
- LYT-300 (Experimental)
  Interventions: Drug: LYT-300
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LYT-300 — A prodrug of allopregnanolone, a small molecule drug
  Arms: LYT-300; LYT-300 in healthy volunteers LYT-300; LYT-300 in healthy volunteers LYT-300, Dose TBD QHS every 24 h for 7 days; LYT-300 in healthy volunteers LYT-300, Doses TBD; LYT-300, Dose TBD QAM every 24 h for 7 days; Placebo QHS every 24 h for 7 days
Other: Placebo — Placebo for LYT-300
  Arms: LYT-300 in healthy volunteers LYT-300, Dose TBD QHS every 24 h for 7 days; LYT-300 in healthy volunteers LYT-300, Doses TBD; Placebo; Placebo QAM every 24 h for 7 days; Placebo QHS every 24 h for 7 days

SUMMARY:
Part 1 is a single ascending dose (SAD) trial in healthy volunteers (HV) to assess the safety, tolerability, and pharmacokinetic (PK) profile of orally administered LYT-300.

Part 2 is a crossover assessment in HV of the effects of food on the safety, tolerability, and PK profile of orally administered LYT-300.

Part 3 is a multiple ascending dose (MAD) trial in HV to assess the safety, tolerability, and PK profile of multiple doses (up to 7 days) of orally administered LYT-300.

Part 4 is an assessment of the effects of LYT-300 vs. placebo on pharmacodynamic and patient reported outcome response to a validated clinical model of anxiety.

DETAILED DESCRIPTION:
Part 1: This is a randomized, double-blind, placebo-controlled, SAD design to assess the safety, tolerability, and PK profile of orally administered LYT-300 in HV, in a 3-period, 3-sequence, crossover, dose escalation design.

Part 2: This is a randomized, open label, 3-period, 3-sequence, crossover assessment of the effects of food on the PK, safety, and tolerability of orally administered LYT-300 in HV. A single dose of LYT-300 will be administered on 3 occasions, separated by a minimum 7-day washout period. Part 2 is planned as a single dosing cohort.

Part 3: This is a randomized, double-blind, placebo-controlled, sequential, MAD trial in HV to assess the safety, tolerability, and PK profile of multiple doses (up to 7 days) of orally administered LYT-300. This part will include ascending doses given either once daily in the morning (QAM), once daily in the evening (QHS), or twice daily (BID).

Part 4: This is a double-blind, randomized assessment of the effects in HV of a single dose of LYT-300 vs. placebo on pharmacodynamic and patient reported outcome response to a validated clinical model of anxiety.

ELIGIBILITY:
Main Inclusion Criteria:

Parts 1, 2, 3 and 4: Healthy Volunteers

1. Male or female between 18 and 55 years old (inclusive) at the time of screening.
2. In good general health at screening, free from clinically significant unstable medical, surgical or psychiatric illness, at the discretion of the Investigator.

Main Exclusion Criteria:

Parts 1, 2, 3 and 4: Healthy Volunteers

1. Evidence or history of any condition or situation that adversely impacts a normal sleep-wake cycle.
2. Confirmed COVID-19 infection within 2 months of screening, known exposure to another person with COVID-19 within 14 days of screening
3. History of illness with fever within 28 days prior to the first dose.
4. A history of, or current evidence for, serious mental illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: treatment-emergent adverse events [TEAEs] | 7 days (main time frame)
  Evaluate the safety and tolerability in healthy volunteers following single or multiple oral doses of LYT-300 as measured by TEAEs.
Effect of food in healthy volunteers | 2 days (main time frame)
  Measure concentration of allopregnanolone in blood plasma in fed or fasted subjects administered a single dose of LYT-300
Salivary cortisol | 60 minutes
  Change in salivary cortisol

SECONDARY OUTCOMES:
Use pharmacokinetics to characterize the blood plasma concentration of allopregnanolone after administration of LYT-300 | 7 days (main time frame)
  Measure the blood plasma concentrations of allopregnanolone in healthy volunteers after single and multiple doses of LYT-300 administered up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No